CLINICAL TRIAL: NCT05353192
Title: A Multicenter, Open-label, Single Arm Phase IV Clinical Study to Evaluate the Efficacy and Safety of Recombinant Human Growth Hormone in Children With Achondroplasia
Brief Title: A Study to Evaluate the Efficacy and Safety of Recombinant Human Growth Hormone in Children With Achondroplasia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Children's Hospital of Fudan University (Other); Tongji Hospital (Other); Children's Hospital of Nanjing Medical University (Other); Jiangxi Province Children's Hospital (Other); Chengdu Women's and Children's Central Hospital (Other); Shandong Provincial Hospital (Other Government); Shengjing Hospital (Other); Shanghai Children's Hospital (Other); Children's Hospital of The Capital Institute of Pediatrics (Other); West China Second University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci001-01
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Achondroplasia
Keywords: Achondroplasia
MeSH Terms: conditions — Achondroplasia | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant human growth hormone (Experimental): Recombinant human growth hormone Injection (15IU/5mg/3ml/bottle)；0.05 mg/kg/d by subcutaneous injection for 52 weeks
  Interventions: Drug: Recombinant human growth hormone

INTERVENTIONS:
Drug: Recombinant human growth hormone — Recombinant human growth hormone (15IU/5mg/3ml/bottle)，0.05 mg/kg/d by subcutaneous injection for 52 weeks

SUMMARY:
To Evaluate the Efficacy and Safety of Recombinant Human Growth Hormone in Children with Achondroplasia

ELIGIBILITY:
Inclusion Criteria:

* 2-10 years old;
* In Tanner I stage;
* ACH, documented and confirmed by genetic testing;
* Short stature;
* Ambulatory and able to stand or walk without assistance;
* Parent(s) or guardian(s) consent；
* Had never been treated with growth hormone

Exclusion criteria:

* Short stature condition other than ACH;
* Evidence of growth plate closure (proximal tibia, distal femur);
* Had a fracture of the long bones within 6 months prior to screening;
* Planned or expected bone-related surgery;
* Chronic diseases condition that affect bone metabolism and weight;
* Severe intracranial hypertension

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Annualized Height Velocity (AHV) at Week 52 | week 52
  The change in AHV after 52 weeks treatment

SECONDARY OUTCOMES:
Change From Baseline in AHV | week 4, week 13, week 26, week 39
  Change in AHV at week, week 13, week 26, week 39
Change From Baseline in Height Standard Deviation Score (Ht SDS) | week 4, week 13, week 26, week 39, week 52
  Change From Baseline in Ht SDS at week 4, week 13, week 26, week 39, week 52
Change From Baseline in BMI Standard Deviation Score (BMI SDS) | week 4, week 13, week 26, week 39, week 52
  Change From Baseline in BMI SDS at week 4, week 13, week 26, week 39, week 52
Change From Baseline in Sitting Height/Leg Length ratio Standard Deviation Score (SH/LL SDS) | week 4, week 13, week 26, week 39, week 52
  Change From Baseline in SH/LL SDS at week 4, week 13, week 26, week 39, week 52
Change From Baseline in IGF-1 Standard Deviation Score (IGF -1 SDS) | week 4, week 13, week 26, week 39, week 52
  Change From Baseline in IGF-1 SDS at week 4, week 13, week 26, week 39, week 52
Change From Baseline in IGF-1/IGFBP-3 ratio | week 4, week 13, week 26, week 39, week 52
  Change From Baseline in IGF-1/IGFBP-3 ratio at week 4, week 13, week 26, week 39, week 52
Change From Baseline in Bone Age/Chronological Age ratio (BA/CA) | week 52
  Change From Baseline in BA/CA at week 52

OTHER OUTCOMES:
Change From Baseline in Metabolism-related Proteins | week 13, week 26, week 52
  Change From Baseline in Serum Proteomics at week 13, week 26, week 52

CONTACTS AND LOCATIONS:
Overall Officials: Feihong Luo, Principal Investigator — Children's Hospital of Fudan University; Xiaoping Luo, Principal Investigator — Tongji Hospital; Wei Gu, Principal Investigator — Children's Hospital of Nanjing Medical University; Yu Yang, Principal Investigator — Jiangxi Province Children's Hospital; Xinran Cheng, Principal Investigator — Chengdu Women's and Children's Central Hospital; Guimei Li, Principal Investigator — Shandong Provincial Hospital; Ying Xin, Principal Investigator — Shengjing Hospital of China Medical Hospital; Pin Li, Principal Investigator — Shanghai Children's Hospital; Xiaobo Chen, Principal Investigator — Children's Hospital of The Capital Institute of Pediatrics; Jin Wu, Principal Investigator — West China Second University Hospital
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Drugs belong to the sponsor before they are put into clinical trials and the site is only a contract research organization; It is an industry practice that intellectual property rights belong to the sponsor.